CLINICAL TRIAL: NCT04479605
Title: Values and Options in Cancer Care 2.0 (VOICE 2.0): Building on Lessons Learned to Improve Communication and Illness Understanding in Cancer Patients and Their Caregivers
Brief Title: Communication Training for Cancer Patients, Their Caregivers, and Their Doctors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-241
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Communication and Illness Understanding
Keywords: Caregiver Support Sessions; Patient & Caregiver Coaching; 20-241
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with advanced cancer: Patient and caregiver coaching is facilitated by a booklet titled Our Cancer Care (Appendices E & F) that includes a Question Prompt List (QPL) and resources for a Values Affirmation Exercise (Appendices G & H). The QPL and Values Affirmation Exercises will be provided with a cover letter (Appendix I). The QPL consists of example questions to discuss with oncologists about diagnosis, prognosis, treatments, symptom management, transitions in care, self-care, family needs, and life goals. Patients and caregivers meet over video-conferencing with a study interventionist for one hour to review the QPL. The interventionist makes three follow-up phone calls to each dyad bi-weekly to evaluate use of the QPL.
- Caregivers: Caregivers will participate in three 45-minute sessions with the interventionist over the telephone or video-conferencing (per caregiver preference) approximately bi-weekly. These sessions take place while the patient and caregiver are completing the three follow-up dyadic sessions. Efforts will be made to schedule the caregiver support sessions during weeks that fall between dyadic coaching sessions to minimize intervention burden on caregivers (i.e., avoiding scheduling two sessions for the caregiver in the same week).
- Oncologists: The Oncologist training will be conducted online using Bridge, an internet-based platform designed to facilitate communication between instructors and learners. The training includes written information on and videos demonstrating target communication skills (Table 1) and knowledge acquisition checks. Five of the online modules are required and the remaining six modules are optional. The required modules are estimated to take oncologists approximately one hour to complete; the optional modules are estimated to take 90 minutes total (i.e., for all modules) to complete. Oncologists' logging history will be tracked in Bridge.

SUMMARY:
The purpose of this study is to develop and test a new communication intervention, "Values and Options in Cancer Care 2.0" (VOICE 2.0), which involves oncologist training, patient and caregiver coaching, and caregiver support.

The VOICE 2.0 intervention was developed by members of the study team to improve communication among oncologists, patients with cancer, and caregivers. Researchers have found that clear communication about the patient's disease can help with the planning of that patient's future care and improve the well-being of both the patient and his or her caregiver. The long-term goals of developing and testing VOICE 2.0 include improving the care and respecting the wishes of cancer patients, and helping those patients and their caregivers have an improved quality of life during their experience with cancer.

ELIGIBILITY:
Inclusion Criteria:

ONCOLOGISTS:

* As per self-report, medical oncologist providing care to patients with gastrointestinal, genitourinary, gynecologic, lung, or hematologic cancers at MSK
* As per self-report, not planning to leave MSK in the next six months
* As per self-report, willing to be audio-recorded for Post-Training Follow-Up Interview

PATIENTS:

* Per medical record and/or self-report, a patient of an oncologist participating in this study
* As per medical record and/or self-report, diagnosis of:

  * a hematologic cancer with disease progression following second-line treatment that is not eligible for transplant; OR
  * stage III or IV gastrointestinal, genitourinary, gynecologic, or lung cancer
* As per medical record and/or self-report, fluent in English
* As per medical record and/or self-report, age 18 or older
* As per self-report, has a primary informal caregiver (as defined by an unpaid individual who provides the patient with emotional, physical, and/or practical support) who is willing and able to participate in the study
* As per self-report, residency in New York or ability to complete sessions in New York to ensure that provision of intervention is covered by the professional licenses of interventionists (i.e., social workers licensed in New York State)
* As per self-report, able to communicate over video-conference and phone for sessions
* As per self-report, willing to be audio-recorded for assessments and study sess

CAREGIVERS:

* As per patient report, is a primary informal caregiver ("a family member, partner, friend, or other individual involved with your health care issues, preferably someone who comes to physician appointments with you") for an MSK patient
* As per self-report, fluent in English
* As per self-report, age 18 or older
* As per self-report, ability to complete sessions in a state the interventionists are legally allowed to practice in (i.e., social workers licensed in New York or New Jersey State; states with shared license laws)
* As per self-report, able to communicate over video-conference and phone for sessions
* As per self-report, willing to be audio-recorded for assessments and study sessions ** Language verification: For both patients and caregivers, prior to enrollment, all will be asked the following two questions by an CRC to verify English fluency necessary for participation in the study:

  1. How well do you speak English? (must respond "Very well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
  2. What is your preferred language for healthcare? (must respond English)

Exclusion Criteria:

PATIENTS:

* Score >4 on Short Portable Mental Status Questionnaire
* As per self-report, feels too weak or cognitively impaired to participate in the intervention and complete the assessments
* As per medical record or self-report, receiving hospice care at the time of enrollment

CAREGIVERS:

* Score >4 on Short Portable Mental Status Questionnaire
* As per self-report, feels too weak or cognitively impaired to participate in the intervention and complete the assessments
* As per medical record or self-report, receiving hospice care at the time of enrollment
* As per patient or self-report, supports the patient in a professional role

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Voice 2.0 consists of Oncologist training, patient and caregiver coaching, and caregiver support.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Feasibility will be assessed by rates of accrual, retention, and intervention completion | 10 weeks
Intervention Acceptability | 7 weeks
  Intervention Acceptability will be assessed with Likert scale items with responses that range from 1 to 5 with higher scores indicating greater acceptability.

SECONDARY OUTCOMES:
Concordant illness understanding (oncologists, patients, caregivers) | 7 weeks
  will be measured using two items assessing participants' beliefs about the patient's chances of living two or more years and chances of being cured. Items are rated on a seven-point scale: 100%, 90% 75%, 50-50, 25%, 10%, 0%. Patient, caregiver, and oncologist responses that differ by two or more response categories will be categorized as discordant.
Communicational self-efficacy | 7 weeks
  will be measured with the 10-item Perceived Efficacy in Patient-Physician Interactions (PEPPI) survey.
Patient-caregiver communication quality | 7 weeks
  will be assessed with the 5-item Family Communication subscale of the Cancer Communication Assessment Tool for Patients and Families, a valid measure in cancer patients and caregivers.
Patient/caregiver-oncologist relationship strength | 7 weeks
  will be measured with the 16-item Human Connection scale Each item is rated on Likert scale from 1 to 4 with higher scores indicating a stronger relationship with the oncologist.
Psychological distress | 7 weeks
  will be measured using the Hospital Anxiety and Depression Scale (HADS), a 14-item self-report measure45 commonly used with cancer patients46-51 and caregivers
Meaning and purpose (patients, caregivers) | 7 weeks
  will be assessed with the 48-item Life Attitude Profile-Revised, a self-report measure of discovered meaning and the motivation to find purpose that has been used with advanced cancer patients and caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Trevino, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT04479605/ICF_000.pdf